CLINICAL TRIAL: NCT03470740
Title: Effects of a Rheumatoid Arthritis Self-management program-a Randomized Controlled Trial
Brief Title: Effects of a Rheumatoid Arthritis Self-management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ChangGungMHRA
Record Dates: First submitted 2018-03-08; First posted 2018-03-20 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2018-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: rheumatoid arthritis, self-management, self-efficacy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to experimental group who received a rheumatoid arthritis self-management intervention based on self-efficacy theory for 6 weeks, and a control group receiving standard rheumatology care only.
Who Masked: Outcomes Assessor
Masking Description: The researcher who collected the data and the researcher who applied the intervention program was never the same.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Other): An individualized rheumatoid arthritis self-management program for managing RA patients' physical behavioral problems was applied for the intervention group. The program was based on the self-efficacy theory and the four resources were incorporated to emphasize patients' knowledge, skill, and responsibility in managing their RA situations.
  Interventions: Behavioral: rheumatoid arthritis self-management program
- control group (No Intervention): The control group received general information on rheumatoid arthritis care and follow-up.

INTERVENTIONS:
Behavioral: rheumatoid arthritis self-management program — The intervention group received the rheumatoid arthritis self-management program which was based on Bandura's theory of self-efficacy and proposes that self-efficacy is influenced by four information sources: mastery of experience, social modeling, social persuasion and one's physical and emotional states. To enhance participants' self-management skill, the following strategies were employed: peer story-telling, assessment, family involvement, goal setting, self-monitoring, self-evaluation, and phone calls consultation.
  Arms: intervention group

SUMMARY:
Rheumatoid arthritis (RA) is a persistent systemic disease. WHO (World Health Organization) commented that a crucial goal of heath care for RA is prevention of loss of daily function by patients' self-management (SM) skills; however, a comprehensive rheumatoid arthritis self-management (RASm) for RA patients' day-to-day self-managing is limited in Taiwan.

Aims: The aims of the study are: (1) to implement the RASm program, (2) to determine the effectiveness of the program with 6 months follow-up, and (3) to understand participants' experiences when receiving the RASm program for the experimental group.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a persistent systemic disease. WHO (World Health Organization) commented that a crucial goal of heath care for RA is prevention of loss of daily function by patients' self-management (SM) skills; however, a comprehensive rheumatoid arthritis self-management program for RA patients' day-to-day self-managing is limited in Taiwan. The aims of the study are: (1) to implement the rheumatoid arthritis self-management program, and (2) to determine the effectiveness of the program with 6 months follow-up. The project will design to implement and evaluate the rheumatoid arthritis self-management program for RA patients using two groups experimental design. A medical center in northern Taiwan will be selected and patients who visited the RA departments will be eligible for the study if they are: (1) diagnosed with RA, (2) age of 20 years or over, (3) disease considered have been stable for at least 3 months, and (4) able to understand and comply with the study treatment. After completion of baseline data, patients will be randomly allocated to the intervention or control group using a computerized allocation procedure and follow the CONSORT flow diagram. Control patients received usual care, and the intervention group will receive the 6-week rheumatoid arthritis self-management program which based on self-efficacy theory. The independent variable of the program will be the four information include mastery experience, social modeling, social persuasion and physical and emotional states, and the strategies involve education, goal setting and attainment, self-monitoring, and phone calls. All participants will follow up for 6 months, and the data will be collected at the baseline, and 2, 3, and 6 months. The statistics with the GEE (generalized estimating equation) analysis will be used to evaluate the outcomes such as the disease activity (DAS-28), arthritis self-efficacy (ASE), physical functioning (MHAQ), quality of life (SF-36), and self-management behaviors. Through enhance the capacity of self-management program for the RA cases to reduce the health care utilization and patients' and caregivers' burden.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA
* Age of 20 years or over
* Disease considered have been stable for at least 3 months
* Able to understand and comply with the study treatment

Exclusion Criteria:

* Suffering from other terminal illnesses, severe dementia or another debilitating psychiatric disorder
* Living in a long-term care facility
* Participation in another research protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Su-Hui Chen, PhD, Principal Investigator — Professor, School of Nursing, Chang Gung University of Science and Technology
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: An individualized home-based rheumatoid arthritis self-management program for managing RA patients' physical behavioral problems was applied for the intervention group. The program was based on the self-efficacy theory and the four resources were incorporated to emphasize patients' knowledge, skill, and responsibility in managing their RA situations.
  rheumatoid arthritis self-management program: The intervention group received the rheumatoid arthritis self-management program which was based on Bandura's theory of self-efficacy and proposes that self-efficacy is influenced by four information sources: mastery of experience, social modeling, social persuasion and one's physical and emotional states. To enhance participants' self-management skill, the following strategies were employed: peer story-telling, assessment, family involvement, goal setting, self-monitoring, self-evaluation, and phone calls consultation.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 112 | 112
Completed | 108 | 106
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.20 (11.29) | 59.47 (11.86) | 58.83 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 98 | 192
  Male | 18 | 14 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 112 | 112 | 224
Duration of RA [Mean (Standard Deviation); unit: years] | 10.21 (8.09) | 11.12 (8.92) | 10.66 (8.51)

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity
Description: Disease activity was measured using the DAS-28 (Disease Activity Score-28) which evaluated 28 tender and swollen joint counts of rheumatoid arthritis patients. This scale was used to calculate the 28 tender and swollen joint counts. Scores can range from 0 to 9.4. The lower score represent a better RA outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 112 | 112
score on a scale | 3.38 (1.15) | 3.62 (1.26)

2. Secondary Outcome: Arthritis Self-efficacy- Pain
Description: We used the arthritis self-efficacy-pain (ASE-pain) to measure RA patients' pain self-efficacy. The ASE-pain used visual analogue scales (0-10), in which 0 means 'very uncertain' and 10 means 'very certain'; a higher score refers to higher self-efficacy. This scale have 5 items, therefore, the score range will be 0-50.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 112 | 112
score on a scale | 35.21 (8.86) | 32.72 (11.16)

3. Secondary Outcome: Arthritis Self-efficacy- Other
Description: We used the arthritis self-efficacy-other (ASE-OS) to measure RA patients' other symptoms self-efficacy. The ASE-OS used visual analogue scales (0-10), in which 0 means 'very uncertain' and 10 means 'very certain'; a higher score refers to higher self-efficacy. This scale have 6 items, therefore, the score range will be 0-60.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 112 | 112
score on a scale | 51.71 (8.98) | 48.96 (11.88)

4. Secondary Outcome: SF-36 Quality of life_Physical Component Scores
Description: The Short-form 36 includes one multi-item scale that assesses 8 dimensions of health: physical functioning (PF), social functioning (SF), role limitations because of physical health problems (RP), bodily pain (BP), general mental health (psychological distress and well-being; MH), limitations in usual role activities because of emotional problems (RE), vitality (energy and fatigue; VT), and general health perceptions (GH), was used to assess the quality of life in this study. The original scale using the Likert scoring method, the score is from 1-3 or 1-5. Before the scores are added, we follow the SF-36 manual, adjust each item scored from 0 to 100, with 0 indicating extreme problems and 100 indicating no problems. The physical component scores (PCS) included GH, PF, RP, and BP, then the scores of each sub-question under the Physical Component Scores are summed together, and the range after adjustment from 0 (extreme problems) to 400 (no problems) for the Physical Component Scores.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 112 | 112
score on a scale | 51.29 (8.72) | 48.88 (10.23)

5. Secondary Outcome: Physical Functioning
Description: The 8-item Modified Health Assessment Questionnaire was used to measure the physical functioning for this study. The MHAQ measures eight activities such as dressing and grooming, arising, eating, walking, hygiene, reach grip, and common daily activities. Items are rated from 1 = without difficulty, to 4 = unable to do; a lower score indicates a greater ability to conduct daily activities. The range of the score will be 8-32.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 112 | 112
score on a scale | 23.72 (7.30) | 26.14 (10.64)

6. Secondary Outcome: Self-management Behaviors
Description: To assess self-management behaviors the researchers developed a joint activity and protection self-management behaviors scale. The scale consists of eight items and ranges from zero for 'never' to four for 'always'. Higher scores indicate a higher level of use of each of the self-management behavior. The range of the score will be 0-32.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 112 | 112
score on a scale | 16.69 (4.80) | 16.24 (4.82)

7. Secondary Outcome: SF-36 Quality of Life_Mental Component Scores (MCS)
Description: The Short-form 36 includes one multi-item scale that assesses 8 dimensions of health: physical functioning (PF), social functioning (SF), role limitations because of physical health problems (RP), bodily pain (BP), general mental health (psychological distress and well-being; MH), limitations in usual role activities because of emotional problems (RE), vitality (energy and fatigue; VT), and general health perceptions (GH), was used to assess the quality of life in this study. The original scale using the Likert scoring method, the score is from 1-3 or 1-5. Before the scores are added, we follow the SF-36 manual, adjust each item scored from 0 to 100, with 0 indicating extreme problems and 100 indicating no problems. The mental component scores (MCS) included RE, SF, VT, and MH, then the scores of each sub-question under the Mental Component Scores are summed together, and the range after adjustment from 0 (extreme problems) to 400 (no problems) for the Mental Component Scores.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 112 | 112
score on a scale | 50.98 (9.36) | 48.97 (10.67)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03470740/Prot_002.pdf
  • Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03470740/SAP_001.pdf